CLINICAL TRIAL: NCT02006511
Title: Incisional Negative Pressure Dressing on Clean Closed Groin Incisions in High Risk Patients
Brief Title: Incisional Negative Pressure Dressing on Clean Closed Groin Incisions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never performed and closed.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00057511
Record Dates: First submitted 2013-11-13; First posted 2013-12-10 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2017-12

CONDITIONS: Complication of Surgical Procedure
Keywords: incisional negative pressure wound therapy; groin incision; incisional VAC; Prevena; groin wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Incisional Neg Pressure Wound Therapy (Experimental): Incisional negative pressure wound therapy dressings applied to the surgical site
  Interventions: Device: Incisional Neg Pressure Wound Therapy (Prevena™)
- Standard of care wound dressing (Active Comparator): Standard of care wound dressing of gauze and tape or the equivalent applied to the surgical site
  Interventions: Other: Standard of Care wound therapy

INTERVENTIONS:
Device: Incisional Neg Pressure Wound Therapy (Prevena™) — Negative pressure wound therapy dressing applied over closed surgical incision
  Arms: Incisional Neg Pressure Wound Therapy
Other: Standard of Care wound therapy — Gauze type dressing.
  Arms: Standard of care wound dressing

SUMMARY:
Wound complications associated with surgical incisions range from minor to life threatening. Surgical site infections occurring usually occur within 30 days and are one of the most common surgical complications. Perigraft infections in groin wounds can be devastating. Even superficial wounds can progress to deep wounds resulting in graft infection, need for explantation, and sepsis or amputation requirement. Negative pressure wound therapy has had favorable results on closed wounds in trauma populations. Similarly, negative pressure wound therapy has had positive benefits in closed incisions such as sternal wounds following cardiac surgery. As a result, the PrevenaTM Incision Management System(IMS) was developed to allow easier application of negative pressure therapy to closed wounds. Application of the PrevenaTM IMS dressing would portend the aforementioned benefits of Vacuum Assisted Closure (VAC®) therapy with the added benefits of protecting the wound from contamination and bolstering the wound edges for better approximation and consequently better aesthetic outcome. However, no comparison between negative pressure therapy as a dressing and standard wound dressings exists.

The purpose of this study is to assess the efficacy and safety of topical negative pressure therapy application with Prevena™ versus standard of care wound therapy on closed groin incisions in high risk patients undergoing vascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or greater
* Scheduled elective vascular surgery which requires groin incision. Elective surgery is defined as planned surgery a minimum of 24 hours before the procedure.
* Meets high risk criteria according to the following rating system
* Scores at least 8 points for the following risk factors:

  • MAJOR 4 points:
* BMI of <18 kg/m2 or ≥BMI 40 kg/m2 ***
* Insulin dependent Diabetes Mellitus*
* Dialysis (hemodialysis or peritoneal dialysis)**

  • INTERMEDIATE 2 points:
* Previous groin surgery
* Diabetes Mellitus not requiring insulin*
* Chronic lung disease GOLD >2
* On long-term immunosuppressive medication (>3 months at time of enrollment)
* Chronic kidney disease (defined as a GFR <30ml/min/1.73m2 for 3 months)**
* Previous lower extremity or abdominal wall radiotherapy radiotherapy
* BMI between 35 and 40***

  • MINOR 1 point:
* Previous abdominal surgery
* Peripheral vascular disease
* Female gender
* Age >75 years old
* Hospitalized at least 7 days before surgery

  *, **, *** mutually exclusive, highest score should be used
* Capable of providing informed consent or has a legally authorized representative (LAR) if unable to provide informed consent
* Willing and able to adhere to the study visit schedule

Exclusion Criteria:

* Subjects meeting any of the following criteria may not be enrolled in the study:
* Is pregnant
* Has a systemic infection at the time of surgery (ie bacteremia)
* Has a remote body site infection at the time of surgery (ie UTI)
* Has a known allergy or hypersensitivity to silver, adhesive, or dressing material
* Has a requirement for competing therapy (ie open negative pressure wound therapy)
* Is simultaneously participating in another interventional trial

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2014-12-01 (Actual)

PRIMARY OUTCOMES:
Deep wound infection | within 30 postoperative days

SECONDARY OUTCOMES:
Superficial Wound Infection | within 30 postoperative days
  Cellulitis or other superficial infection of the wound or tissue immediately surrounding the wound
Wound dehiscence | within 30 postoperative days
  Spontaneous opening of a previously closed surgical wound

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Bluebond-Langer, MD, Principal Investigator — University of Maryland, School of Medicine, Dept of Surgery, Division of Plastic Surgery
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States